CLINICAL TRIAL: NCT02071225
Title: Phase II Trial to Evaluate The Efficacy of Obinutuzumab (RO5072759) + Bendamustine Treatment in Patients With Refractory Or Relapsed Chronic Lymphocytic Leukemia
Brief Title: A Study Evaluating the Efficacy of Obinutuzumab and Bendamustine Treatment in Participants With Refractory or Relapsed Chronic Lymphocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML29167; 2013-003388-79 (EudraCT Number)
Record Dates: First submitted 2014-02-21; First posted 2014-02-25 (Estimated); Results first posted 2019-11-26 (Actual); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Bendamustine Hydrochloride; obinutuzumab

ARMS (1):
- Obinutuzmab + Bendamustine (Experimental): Participants will receive obinutuzumab and bendamustine in 28-days cycles for a maximum of 6 cycles
  Interventions: Drug: bendamustine; Drug: obinutuzumab

INTERVENTIONS:
Drug: bendamustine — 70 milligrams per square meter (mg/m^2) given by intravenous (IV) infusion on Days 2 and 3 of Cycle 1 and on Days 1 and 2 of subsequent cycles.
Drug: obinutuzumab — 1000 mg given by IV infusion on Days 1, 8, and 15 of Cycle 1 and on Day 1 of subsequent cycles.
  Other Names: RO5072759

SUMMARY:
This phase II trial was designed to evaluate the efficacy of obinutuzumab and bendamustine treatment in participants with refractory or relapsed chronic lymphocytic leukemia (CLL). Participants receive up to six 28-day cycles of treatment. Treatment consists of intravenous (IV) administration of obinutuzumab and bendamustine. Treatment time is expected to last 6 months, and participant follow-up will last 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Diagnosed CD20+ B- chronic lymphocytic leukemia (CLL) according to National Cancer Institute (NCI) criteria
* Active disease meeting at least 1 of the International Workshop on CLL (IWCLL) 2008 criteria for treatment
* Refractory CLL (i.e. treatment failure or progression during treatment or within 6 months after the last treatment) or relapse CLL (i.e. participants who met criteria for CR or PR, but progressed beyond 6 months post-treatment)
* At least 1 prior purine analogue or bendamustine containing therapy
* Life expectancy greater than (>) 6 months
* Use of effective contraception as described in the study protocol

Exclusion Criteria:

* Prior Alogenic Bone Marrow Transplant
* Greater than or equal to (>/=) 3 previous lines of chemotherapy and/or immunotherapy for the CLL
* Previous obinutuzumab-containing regimen
* Treatment failure or progression within 6 months of bendamustine-containing regimen
* Transformation of CLL to aggressive non-Hodgkin lymphoma (NHL; Richter's transformation) Patients with prolymphocytic transformation cannot entry the study either
* Active haemolytic anaemia
* Inadequate liver function
* History of other malignancy which could affect compliance with the protocol or interpretation of results. Patients with a history of malignancy that has been treated but not with curative intent will be excluded, unless the malignancy has been in remission without treatment for >/= 2 years prior to enrolment. Patients with a history of adequately treated carcinoma in situ of the cervix; basal or squamous cell skin cancer; low grade, early stage localized prostate cancer treated surgically with curative intent; good prognosis ductal carcinoma in situ (DCIS) of the breast treated with lumpectomy alone with curative intent are eligible
* Evidence of significant, uncontrolled concomitant diseases that could affect compliance with the protocol or interpretation of results, including significant cardiovascular disease or pulmonary disease
* Recent major surgery (within 4 weeks prior to the start of Cycle 1), other than for diagnosis
* Regular treatment with corticosteroids during the 4 weeks prior to study start, unless administered for another condition at a dose equivalent to less than or equal to (</=) 30 milligrams per day (mg/day) prednisone
* Known active infection or any infection requiring treatment with IV antibiotics or hospitalization within 4 weeks prior to study start
* Patients with HIV, human T cell leukemia virus 1 (HTLV-1), hepatitis B or hepatitis C
* Pregnancy or breast-feeding
* Vaccination with a live vaccine within 4 weeks prior to baseline visit
* Receipt of any other study drug within 4 weeks prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2014-04-09 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Spain (21):
  - Hospital De Txagorritxu; Servicio de Hematologia, Vitoria-Gasteiz, Alava
  - Hospital General Universitario de Elche; Servicio de Hematologia, Elche, Alicante
  - Hospital Universitari Germans Trias i Pujol; Servicio de Hematologia, Badalona, Barcelona
  - Hospital Mutua de Terrassa; Servicio de Hematologia, Terrassa, Barcelona
  - Hospital General de Castellon; Servicio de Hematologia, Castellon, Castellon
  - Hospital de Navarra, Servicio de Hematología, Pamplona, Navarre
  - Hospital de Cabueñes; Servicio de Hematología y Hemoterapia, Gijón, Principality of Asturias
  - Hospital Univ. Central de Asturias; servicio de Hematologia, Oviedo, Principality of Asturias
  - Complejo Hospitalario Nuestra Señora de la Candelaria; Servicio de Hematologia, Santa Cruz de Tenerife, Tenerife
  - Hospital Universitari Vall d'Hebron; Servicio de Hematologia, Barcelona
  - Hospital Clínic i Provincial; Servicio de Hematología y Oncología, Barcelona
  - Hospital Universitario Virgen de las Nieves; Servicio de Hematologia, Granada
  - Hospital de Gran Canaria Dr. Negrin; Servicio de Hematologia, Las Palmas
  - Hospital Universitario la Paz; Servicio de Hematologia, Madrid
  - Hospital Universitario Puerta de Hierro; Servicio de Hematologia, Madrid
  - Hospital Costa del Sol; Servicio de Hematologia, Málaga
  - Hospital Universitario Virgen Macarena; Servicio de Hematologia, Seville
  - Hospital Univ. Nuestra Señora de Valme; Servicio de Hematologia, Seville
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia
  - Hospital Universitario Dr. Peset; Servicio de Hematologia, Valencia
  - Hospital Clinico Universitario Lozano Blesa; Servicio de Hematologia, Zaragoza

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 72 participants were recruited at 20 sites in Spain.
Pre-assignment Details: Participants enrolled in the study had documented CD20-positive B-cell type relapsed or refractory chronic lymphocytic leukemia (CLL).
Groups:
- Obinutuzumab + Bendamustine: Participants received obinutuzumab and bendamustine in 28-days cycles for a maximum of 6 cycles.
Period: Overall Study
Arm/Group | Obinutuzumab + Bendamustine
Started | 72
Completed | 42
Not Completed | 30
Not completed — Withdrawal of Consent | 2
Not completed — Protocol Deviation | 1
Not completed — Lost to Follow-up | 2
Not completed — Death | 25

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants, who received at least one dose of any treatment.
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 72
Age, Continuous [Median (Full Range); unit: years] | 67.9 [42.5 to 83.1]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 48
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 71
  Indian | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Assessed by the Investigator Using the International Workshop on Chronic Lymphocytic Leukemia (IWCLL) 2008 Criteria
Description: ORR was defined as percentage of participants achieving Complete Response (CR), incomplete CR (CRi) or Partial Response (PR). CR: lymphocytes below 4 x 10^9/L, absence of lymphadenopathy, hepatomegaly and splenomegaly, absence of disease or constitutional symptoms, neutrophils > 1.5 x 10^9/L, platelets > 100 x 10^9/L, hemoglobin > 110 g/L, bone marrow at least normocellular for age. CRi: CR with persistent cytopenia, i.e. anemia, thrombocytopenia and/or neutropenia. PR: reduction ≥ 50% of the lymphocyte count AND reduction ≥ 50% of the lymphadenopathy OR reduction ≥ 50% of the size of the liver if enlarged at baseline OR reduction ≥ 50% of the size of the spleen if enlarged at baseline PLUS one of the following: neutrophils > 1.5 x 10^9/L, platelets > 100 x 10^9/L, hemoglobin > 110 g/L or increase ≥ 50% compared to pre-treatment.
Time Frame: 2-3 months after last dose of the study treatment (up to approximately 9 months)
Population: Efficacy population included all participants, who received at least one dose of both treatments (bendamustine and obinutuzumab).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 70
percentage of participants | 78.6 [66.8 to 87.1]

2. Secondary Outcome: Best Response Rate as Assessed by the Investigator Using the IWCLL 2008 Criteria
Description: Best overall response was defined as percentage of participants achieving a best response of CR, CRi and PR. CR: lymphocytes below 4 x 10^9/L, absence of lymphadenopathy, hepatomegaly and splenomegaly, absence of disease or constitutional symptoms, neutrophils > 1.5 x 10^9/L, platelets > 100 x 10^9/L, hemoglobin > 110 g/L, bone marrow at least normocellular for age. CRi: CR with persistent cytopenia, i.e. anemia, thrombocytopenia and/or neutropenia. PR: reduction ≥ 50% of the lymphocyte count AND reduction ≥ 50% of the lymphadenopathy OR reduction ≥ 50% of the size of the liver if enlarged at baseline OR reduction ≥ 50% of the size of the spleen if enlarged at baseline PLUS one of the following: neutrophils > 1.5 x 10^9/L, platelets > 100 x 10^9/L, hemoglobin > 110 g/L or increase ≥ 50% compared to pre-treatment.
Time Frame: During study treatment and until 6 months after end of study treatment at approximately 12 months
Population: Efficacy population included all participants, who received at least one dose of both treatments (bendamustine and obinutuzumab). Reported here is the number of participants for whom data for best response achieved were available.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 54
percentage of participants
  CR | 46.3
  CRi | 1.9
  PR | 42.6

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the start of treatment to disease progression (DP), relapse or death from any cause, whichever occurs first, as assessed by the investigator. DP: at least one of the following characteristics: increase ≥ 50% in lymphocytes up to at least 5 x 10^9/L, appearance of new palpable lymph nodes, increase ≥ 50% of the longest diameter of any previous area of clinically significant lymphadenopathy, increase ≥ 50% of the size of the liver and/or spleen, transformation to a more aggressive histology, after treatment progression of any cytopenia: decrease of hemoglobin levels of more than 20 g/L or to below 100 g/L and/or decrease of platelet counts by more than 50% or to below 100 x 10^9/L and/or decrease in the neutrophil counts by more than 50% or to below 1.0 x 10^9/L if the marrow biopsy also shows infiltration of clonal chronic lymphocytic leukemia (CLL) cells.
Time Frame: From start of treatment up to disease progression or relapse or death, whichever occurred first (up to approximately 4.5 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 70
months | 24.14 [20.81 to 27.47]

4. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the start of study treatment to death from any cause.
Time Frame: From start of treatment up to death of any cause (up to approximately 4.5 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 70
months | NA [NA to NA] — Median of OS for efficacy population was not reached.

5. Secondary Outcome: Event Free Survival (EFS)
Description: EFS was defined as the time from the start of treatment to DP/relapse, death from any cause or start of a new anti-leukemia therapy. DP: at least one of the following characteristics: increase ≥ 50% in lymphocytes up to at least 5 x 10^9/L, appearance of new palpable lymph nodes, increase ≥ 50% of the longest diameter of any previous area of clinically significant lymphadenopathy, increase ≥ 50% of the size of the liver and/or spleen, transformation to a more aggressive histology, after treatment, progression of any cytopenia: decrease of hemoglobin levels of more than 20 g/L or to below 100 g/L and/or decrease of platelet counts by more than 50% or to below 100 x 10^9/L and/or decrease in the neutrophil counts by more than 50% or to below 1.0 x 10^9/L if the marrow biopsy also shows infiltration of clonal CLL cells.
Time Frame: From start of treatment up to disease progression or relapse or death or start of a new anti-leukemic therapy, whichever occurred first (up to approximately 4.5 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 70
months | 24.14 [19.96 to 28.32]

6. Secondary Outcome: Disease Free Survival (DFS)
Description: DFS was defined for all participants who achieved complete response (CRi or CR). DFS lasted from the date on which CRi or CR was recorded until the date on which the first DP or death from any cause occurred. DP: at least one of the following characteristics: increase ≥ 50% in lymphocytes up to at least 5 x 10^9/L, appearance of new palpable lymph nodes, increase ≥ 50% of the longest diameter of any previous area of clinically significant lymphadenopathy, increase ≥ 50% of the size of the liver and/or spleen, transformation to a more aggressive histology, after treatment, progression of any cytopenia: decrease of hemoglobin levels of more than 20 g/L or to below 100 g/L and/or decrease of platelet counts by more than 50% or to below 100 x 10^9/L and/or decrease in the neutrophil counts by more than 50% or to below 1.0 x 10^9/L if the marrow biopsy also shows infiltration of clonal CLL cells.
Time Frame: From occurrence of complete response up to disease progression or death, whichever occurred first (up to approximately 4.5 years)
Population: Efficacy population included all participants, who received at least one dose of both treatments (bendamustine and obinutuzumab). Included in the analysis are participants who achieved CRi or CR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 25
months | 23.02 [21.38 to 24.66]

7. Secondary Outcome: Duration of Response (DR)
Description: DR was defined for participants with CRi, CR or PR. DR spanned from the date on which response was recorded until the date on which DP or death from any cause occurred. DP: at least one of the following characteristics: increase ≥ 50% in lymphocytes up to at least 5 x 10^9/L, appearance of new palpable lymph nodes, increase ≥ 50% of the longest diameter of any previous area of clinically significant lymphadenopathy, increase ≥ 50% of the size of the liver and/or spleen, transformation to a more aggressive histology, after treatment, progression of any cytopenia: decrease of hemoglobin levels of more than 20 g/L or to below 100 g/L and/or decrease of platelet counts by more than 50% or to below 100 x 10^9/L and/or decrease in the neutrophil counts by more than 50% or to below 1.0 x 10^9/L if the marrow biopsy also shows infiltration of clonal CLL cells.
Time Frame: From occurrence of CR or PR up to disease progression or death, whichever occurred first (up to approximately 4.5 years)
Population: Efficacy population included all participants, who received at least one dose of both treatments (bendamustine and obinutuzumab). Included in the analysis are participants who achieved CRi, CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 54
months | 21.41 [17.60 to 25.22]

8. Secondary Outcome: Time to Re-treatment/New Anti-leukemia Therapy
Description: Time to re-treatment/new leukemia therapy was defined as the time between the start of treatment and the date of the first administration of re-treatment or new leukemia therapy.
Time Frame: Up to 4.5 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 70
months | NA [NA to NA] — Median of time to re-treatment for efficacy population was not reached.

9. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Negativity
Description: MRD negativity was defined as the presence of less than 1 cell of CLL per 10,000 leukocytes (= category 0, <0.01%) assessed in bone marrow (BM) and peripheral blood (PB) by flow cytometry after the end of the treatment at the final response assessment.
Time Frame: At approximately 9 months
Population: ITT population included all participants, who received at least one dose of any treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 72
percentage of participants
  MRD in BM: Cat 0 | 36.4
  MRD in PB: Cat 0 | 53.4

10. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as AEs. An SAE was any AE that was any of the following: fatal, life-threatening, required or prolonged inpatient hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/ birth defect, and was considered a significant medical event by the investigator.
Time Frame: Up to approximately 4.5 years
Population: Safety population included all participants, who received at least one dose of any treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 72
percentage of participants
  AEs | 94.4
  SAEs | 51.4

11. Secondary Outcome: Percentage of Participants With AEs of Special Interest (AESIs)
Description: AESIs included any of the following: SAEs associated with the infusion of obinutuzumab: obinutuzumab serious infusion-related reactions, which were defined as AEs occurring during or within 24 hours following the administration of an infusion of obinutuzumab and considered related to obinutuzumab; serious infection; serious neutropenia; any tumor lysis syndrome (TLS); second malignancies.
Time Frame: Up to approximately 4.5 years
Population: Safety population included all participants, who received at least one dose of any treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 72
percentage of participants | 45.8

12. Secondary Outcome: Percentage of Participants With Infusion-related Reactions (IRRs)
Description: IRRs were defined as AEs occurring during or within 24 hours following the administration of an infusion and considered related to drug treatment.
Time Frame: Up to end of treatment at 6 months
Population: Safety population included all participants, who received at least one dose of any treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 72
percentage of participants | 20.8

13. Secondary Outcome: Percentage of Participants Who Discontinued Treatment Prematurely
Time Frame: Up to end of treatment at 6 months
Population: Safety population included all participants, who received at least one dose of any treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 72
percentage of participants | 41.7

14. Secondary Outcome: Percentage of Participants With Previous/Concomitant Diseases
Time Frame: Up to approximately 4.5 years
Population: Safety population included all participants, who received at least one dose of any treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 72
percentage of participants | 97.2

15. Secondary Outcome: Percentage of Participants With Concomitant Medication
Description: Concomitant therapies included any medication (prescription medication, over-the-counter medications, herbal/homeopathic remedies, nutritional supplements) used by subjects in the 7 days prior to screening until the end of treatment. The following treatments were not permitted during the study treatment period: investigational or unauthorized or unapproved medicinal products, immunotherapy or radioimmunotherapy (other than the trial immunotherapy, obinutuzumab), chemotherapy (other than the trial chemotherapy, bendamustine) and radiotherapy.
Time Frame: From 7 days prior to screening to the end of treatment at 6 months
Population: Safety population included all participants, who received at least one dose of any treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Obinutuzumab + Bendamustine
Number analyzed (Participants) | 72
percentage of participants | 54.2

ADVERSE EVENTS:
Time Frame: Up to approximately 4.5 years
Description: Safety population included all participants, who received at least one dose of any treatment.
Arm/Group | Obinutuzumab + Bendamustine
All-Cause Mortality (participants affected / at risk) | 25/72
Serious Adverse Events (participants affected / at risk) | 37/72
Other Adverse Events (participants affected / at risk) | 67/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + Bendamustine (N=72)
Neutropenia (Blood and lymphatic system disorders) | 9
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Acute myeloid leukaemia (Blood and lymphatic system disorders) | 1
Acute myelomonocytic leukaemia (Blood and lymphatic system disorders) | 1
Haemophagocytic lymphohistiocytosis (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Dyspnoea (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Gastroenteritis (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Pyrexia (General disorders) | 8
Infusion related reaction (General disorders) | 2
Multiple organ dysfunction syndrome (General disorders) | 2
Cachexia (General disorders) | 1
Malaise (General disorders) | 1
Mucosal inflammation (General disorders) | 1
Pneumonia (Infections and infestations) | 8
Respiratory tract infection (Infections and infestations) | 6
Septic shock (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Abdominal Sepsis (Infections and infestations) | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Periorbital cellulitis (Infections and infestations) | 1
Respiratory syncytial virus infection (Infections and infestations) | 1
Rotavirus infection (Infections and infestations) | 1
Serratia sepsis (Infections and infestations) | 1
Tuberculosis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Gastrointestinal stromal tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Laryngeal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bronchiolitis (Respiratory, thoracic and mediastinal disorders) | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypertensive crisis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Obinutuzumab + Bendamustine (N=72)
Neutropenia (Blood and lymphatic system disorders) | 48
Thrombocytopenia (Blood and lymphatic system disorders) | 30
Anaemia (Blood and lymphatic system disorders) | 14
Dyspnoea (Cardiac disorders) | 6
Chest pain (Cardiac disorders) | 4
Nausea (Gastrointestinal disorders) | 17
Diarrhoea (Gastrointestinal disorders) | 16
Constipation (Gastrointestinal disorders) | 9
Vomiting (Gastrointestinal disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 5
Abdominal pain upper (Gastrointestinal disorders) | 4
Asthenia (General disorders) | 28
Pyrexia (General disorders) | 27
Infusion related reaction (General disorders) | 13
Hypertransaminasaemia (Hepatobiliary disorders) | 4
Respiratory tract infection (Infections and infestations) | 19
Urinary tract infection (Infections and infestations) | 6
Herpes zoster (Infections and infestations) | 5
Decreased appetite (Metabolism and nutrition disorders) | 5
Headache (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 9
Rash (Skin and subcutaneous tissue disorders) | 6
Hypotension (Vascular disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/25/NCT02071225/Prot_SAP_000.pdf